CLINICAL TRIAL: NCT02413970
Title: Inspire® Upper Airway Stimulation System (UAS): Post-Approval Study Protocol Number 2014-001
Brief Title: Inspire® Post-Approval Study / Protocol Number 2014-001
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inspire Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-001
Record Dates: First submitted 2015-03-30; First posted 2015-04-10 (Estimated); Last update posted 2024-12-27 (Actual); Status verified 2024-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSA; Neurostimulation; Hypoglossal nerve; Tongue; Upper airway stimulation; Surgery
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Inspire UAS
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inspire® UAS System (Other): This is a single-arm study; all participants will be implanted with the Inspire® UAS System.
  Interventions: Device: Inspire® UAS System

INTERVENTIONS:
Device: Inspire® UAS System — This is a single-arm study; all participants will be implanted with the Inspire® UAS System, which is a permanent, implantable therapy that consists of three implantable components: an IPG, a stimulation lead, and a sensing lead. In addition, the study subject receives a remote control to activate the therapy.
  Other Names: Inspire® therapy

SUMMARY:
The purpose of this study is to obtain additional long-term safety and efficacy data on the use of Inspire therapy.

DETAILED DESCRIPTION:
This is a multi-center, prospective, single-arm study conducted under a common protocol. Each subject will serve as their own control. Each subject will be followed for 5 years from date of implant.

Potential study subjects will be considered for study participation and consented once pre-implant screening and implant qualification process have been completed. This includes an in-lab PSG, surgical consultation, and a drug-induced sleep endoscopy procedure.

This study will collect pre-operative baseline data including, verification of ineffective CPAP treatment, PSG information, medical history and subject quality of life measures. Intra- and post- operative procedure data will be collected.

Post-implant, procedure- and device-related adverse events, QoL questionnaires, Functional Tongue Exam, therapy usage and device adjustment data will be collected. In-lab PSG sleep study data will be collected during the 2-month and 1 & 3 year follow-up visits, home sleep tests will be conducted and data collected at the 6-month and 2, 4, & 5 year follow-up visits.

The subject population will consist of otherwise healthy men and women that are at least 22 years old and have: 1) Provided written informed consent to participate, 2) Indicated a willingness to comply with the study requirements for the specified follow-up duration, and 3) Met all inclusion and exclusion criteria of this protocol.

Up to 127 subjects will be implanted at a minimum of 10 and a maximum of 20 qualified sites in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Likely suffer moderate-to-severe OSA based on history and physical or have an established diagnosis of OSA (AHI >= 15) based on a prior sleep study
2. Documentation the subject not effectively treated with CPAP therapy. (Examples include non-compliance, discomfort, undesirable side effects, symptoms persist despite use). Subjects who have been prescribed, but refuse to try CPAP would be considered intolerant.
3. Age 22 or above
4. Willing and capable to have stimulation hardware permanently implanted, and to use the patient remote to activate the stimulation
5. Willing and capable to return for all follow-up visits and conduct sleep studies at home, including the evaluation procedures and filling out questionnaires
6. Willing and capable of providing informed consent

Exclusion Criteria:

Contraindications:

1. Central + mixed apneas > 25% of the total apnea-hypopnea index (AHI)
2. Any anatomical finding that would compromise the performance of upper airway stimulation, such as the presence of complete concentric collapse of the soft palate
3. Any condition or procedure that has compromised neurological control of the upper airway
4. Patients who are unable or do not have the necessary assistance to operate the patient remote
5. Patients who are pregnant or plan to become pregnant
6. Patients who will require magnetic resonance imaging (MRI)
7. Patients with an implantable device that may be susceptible to unintended interaction with the Inspire system.

Additional exclusions for study purposes only:

1. Any chronic medical illness or condition that contraindicates a surgical procedure under general anesthesia, as judged by the clinical study Investigator
2. Has a terminal illness with life expectancy < 12 months
3. Active psychiatric disease (psychotic illness, major depression, or acute anxiety attacks) which prevents subject compliance with the requirements of the investigational study testing
4. Any other reason the investigator deems subject is unfit for participation in the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Long-term Device-Related SAEs | 5 Years Post-Implant
  This safety endpoint is to assess long-term (5 years) safety via comparison of device-related SAEs with a performance goal of 24%. The objective at 5 years is to demonstrate the device-related SAE rate is no worse than the performance goal.
Therapy Specific AEs | 12 Months Post-Implant
  This safety endpoint is to evaluate the safety of the Inspire system in the treatment of sleep apnea by evaluating procedure- and device-related AEs occurring immediately post-implant through 12 months post-implant.
Long-term Therapy-Related AEs | 5 Years Post-Implant
  This safety endpoint is to assess long-term (5 years) safety via the description of all reported AEs, including all therapy- and procedure-related events.

SECONDARY OUTCOMES:
Number of Acute AEs Reported with Newly Trained Physicians as Compared to Experienced Physicians | 30 days post-implant
  This endpoint is to assess the performance of newly trained physicians, the post-approval study will collect surgical times, post-operative pain recovery, procedure related AEs, and post-operative comments.

OTHER OUTCOMES:
Change in ESS From Baseline to 12 Months | Baseline and 12 Months
  The Epworth Sleepiness Scale (ESS) is a validated instruction that rates a subject's daytime sleepiness. The ESS efficacy endpoint will be determined by the ESS score at the 12-month follow-up as compared to baseline.
Change in FOSQ From Baseline to 12 Months | Baseline and 12 Months
  The Functional Outcomes of Sleep Questionnaire (FOSQ) is a validated instrument to assess the effect of a subject's daytime sleepiness on activities of ordinary living. The FOSQ endpoint will be determined by the FOSQ score at the 12-month follow-up as compared to baseline.
Change in ODI From Baseline to 3 Years | Baseline and 3 Years
  Oxygen Desaturation Index (ODI) is a measure of OSA severity. The ODI will be determined by the ODI score at the 3-year follow-up compared with the pre-implant baseline score.
Change in AHI From Baseline to 3 Years | Baseline and 3 Years
  Apnea Hypopnea Index (AHI) is a measure of OSA severity. The AHI in this study will be determined by the AHI score at the 3-year follow-up compared with the pre-implant baseline score.

CONTACTS AND LOCATIONS:
Overall Officials: Gwen Gimmestad, Study Director — Inspire Medical Systems, Inc.
Locations (14):
- United States (14):
  - The University of Alabama at Birmingham Medical Center, Birmingham, Alabama
  - University of Southern California, Los Angeles, California
  - South Miami Hospital, Miami, Florida
  - Tampa General Hospital, Tampa, Florida
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Kentucky Research Group, Louisville, Kentucky
  - Weill Cornell Medicine, New York, New York
  - The Christ Hospital, Cincinnati, Ohio
  - University Hospitals, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania, Division of Sleep Medicine, Philadelphia, Pennsylvania
  - Thomas Jefferson University and Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina